CLINICAL TRIAL: NCT04808141
Title: Digital Care Program for Chronic Low Back Pain Versus Conventional Physical Therapy: a Prospective, Randomized Controlled Study
Brief Title: Digital Care Program for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sword Health, SA (Industry)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SH-RCT-LBP-US-01
Record Dates: First submitted 2021-03-12; First posted 2021-03-22 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Outcomes Assessor
Masking Description: Blinding of investigators and patients regarding allocation arm will not be possible, given the nature of the intervention. Analysis of study results will be performed by a statistician blinded to allocation groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Digital Rehabilitation (Experimental): Home-based rehabilitation with a digital biofeedback system
  Interventions: Device: Digital program
- Conventional rehabilitation at an outpatient clinic (Active Comparator)
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Device: Digital program — Patients in the digital intervention group will benefit from an 8-week program composed of therapeutic exercise, education and cognitive behavioural therapy (CBT) program provided by SWORD Health. These patients will be referred to SWORD Health by the investigator who identified the candidate. SWORD Health will then assign a physical therapist to each patient. The physical therapist will contact the patient for onboarding and will manage the case.
  Arms: Digital Rehabilitation
Other: Conventional physical therapy — Patients in this group will benefit from a 8-week program consisting of two 30 min face-to-face physical therapy sessions per week in an outpatient clinic setting, for a total of 16 sessions. The program will follow the protocol outlined in Annex 3, which can however be adapted by the physical therapist to the specific needs of the participant. Participants in this group will be considered as dropouts if they: a) choose to abandon the study; b) miss four consecutive scheduled physical therapy sessions.
  Arms: Conventional rehabilitation at an outpatient clinic

SUMMARY:
New ways of delivering care are much needed to address chronic low back pain. Crucially, these need to: a) address the three pillars of care to achieve good and sustained clinical outcomes; b) overcome barriers to access; c) ensure patients are engaged throughout the programs; d) be scalable and cost-efficient. SWORD Health has developed a digital care program to address these needs. This study aims to assess the clinical outcomes of this rehabilitation program versus conventional physical therapy.

DETAILED DESCRIPTION:
Low back pain (LBP) has for long been the world's leading cause of years leaved with disability,1 and, considering that the overall life expectancy is rising, this pandemic only tends to get worse. Nearly everyone is affected by LBP at some moment in life (70-80% of lifetime prevalence). As a consequence, LBP is also presented as a leading cause of work absenteeism worldwide. Thus, although the estimate costs of LBP may be difficult to compare between different countries, its overwhelming socio-economic impact in modern society is evident.

In the absence of an effective treatment, LBP can become chronic, causing a huge impact in patients' daily life, and ultimately promoting a high consumption of healthcare resources. In the US alone, health expenditures for adults with spinal problems were estimated at $6000 per person, representing a total cost of $102 billion each year.

The dim picture described above highlights the urgent need for effective interventions that minimize disability, improve quality of life and decrease productivity losses.

Current guidelines on CLBP management recommend patient education, exercise, physical therapy (PT), and behavioural therapy as the mainstay treatments for this condition.

Despite some discrepancy in the type of exercise program (e.g. aquatic exercises, stretching, back schools, McKenzie exercise approach, yoga, tai-chi) and mode of delivery (e.g., individually designed programs, supervised home exercise, and group exercise), exercise therapy is recommended nearly transversally, with most studies concluding that exercise intervention programs should include a combination of muscular strength, flexibility and aerobic fitness exercises. Moreover, home exercises with a regular therapist follow-up has proven highly effective.

This is not, however, how LBP is currently managed. Appropriate patient education and structured behavioural training are rarely provided, and opioid prescription is also a common practice, despite known opioid-related morbidity and mortality rates. Because the prevalence of CLBP is continuously rising, and opioid misuse is an issue of great concern globally, identifying effective nonopioid alternatives for CLBP is of paramount importance.

Further compounding this problem, from the patients who are directed to PT, almost half give up after just 4 sessions, and only 30% complete their programs.

In this context, new ways of delivering care are much needed. Crucially, these need to: a) address the three pillars of care to achieve good and sustained clinical outcomes; b) overcome barriers to access; c) ensure patients are engaged throughout the programs; d) be scalable and cost-efficient.

This study aims to assess the clinical outcomes of a digital program for chronic low back pain versus conventional PT.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 80 years of age at enrolment
* Reporting intermittent or persistent low back pain for at least 12 weeks, and/or present at least 50% of the time in the past 6 months
* Ability to understand complex motor tasks

Exclusion Criteria:

* Known pregnancy
* Submitted to spinal surgery less than 3 months ago
* Symptoms and/or signs indicative of possible infectious disorder
* Known disorder with indication for spine surgery (i.e., tumor, cauda equina syndrome)
* Cancer diagnosis or undergoing treatment for cancer
* Cardiac, respiratory or other known disorder incompatible with at least 20 minutes of light to moderate physical activity
* Concomitant neurological disorder (e.g. Stroke, multiple sclerosis, Parkinson's disease)
* Dementia or psychiatric disorders precluding patient from complying with a home-based exercise program
* Illiteracy and/or serious visual or auditory impairment interfering with communication or compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cui Di, MD, Principal Investigator — Emory University
Locations (1):
- Emory Orthopaedic and Spine Center (Atlanta, Ga), Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be made available in PDF format. Aggregate study results, with anonymised individual participant data will be made available in Excel format
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon study publication, for at least five years.
Access Criteria: Study protocol will be made available in clinicaltrials.gov and the excel file with the aggregate results will be made available upon study publication, for at least 5 years.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Started | 70 | 70
Completed | 57 | 45
Not Completed | 13 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50.50 [39.25 to 61.50] | 54.50 [43.00 to 63.25] | 52.00 [40.00 to 63.00]
Age, Customized [Count of Participants; unit: Participants]
  <25 | 1 | 4 | 5
  25-40 | 21 | 10 | 31
  41-60 | 30 | 31 | 61
  >60 | 18 | 25 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 49 | 95
  Male | 24 | 21 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Pacific Islander | 11 | 6 | 17
  Black or African American | 27 | 34 | 61
  Hispanic or Latino | 3 | 2 | 5
  Native American or Alaskan Native | 0 | 1 | 1
  White or Caucasian | 28 | 23 | 51
  Multi-racial or biracial | 0 | 2 | 2
  Prefer not to answer | 1 | 2 | 3
Education level [Count of Participants; unit: Participants]
  Did not attend school | 0 | 1 | 1
  Some high school | 2 | 2 | 4
  High school graduate or GED | 7 | 5 | 12
  Some colleges (some community colleges, associate degree) | 17 | 19 | 36
  Four-year college degree or bachelor's degree | 17 | 14 | 31
  Some postgraduate or professional schooling, no postgraduate degree | 4 | 6 | 10
  Postgraduate or professional degree (including master's, doctorate, medical or law degree) | 23 | 22 | 45
  Prefer not to answer | 0 | 1 | 1
Body Mass Index, categories [Count of Participants; unit: Participants]
  Normal (18.5-25) | 21 | 21 | 42
  Overweight (>25-30) | 21 | 22 | 43
  Obese (>30-40) | 23 | 21 | 44
  Morbidly obese (>40) | 5 | 6 | 11
Employment status [Count of Participants; unit: Participants]
  Employed (part-time or fulltime) | 48 | 46 | 94
  Unemployed (seeking opportunities) | 7 | 4 | 11
  Not employed and not seeking work | 14 | 18 | 32
  Prefer not to answer | 1 | 2 | 3
Exercise levels [Count of Participants; unit: Participants]
  None | 10 | 14 | 24
  Less than 1 h | 20 | 13 | 33
  Between 1-2.5 h | 18 | 24 | 42
  >2.5 h | 22 | 19 | 41
Smoking status [Count of Participants; unit: Participants] — Number of participants who reported being current smokers at baseline measured through the question "Do you smoke?". Participants were classified as smokers or non-smokers based on their responses.
  Participants | 1 | 3 | 4
Low back-related leg pain [Count of Participants; unit: Participants] | 34 | 41 | 75
Laterality of leg pain [Count of Participants; unit: Participants]
  Right | 13 | 16 | 29
  Left | 14 | 13 | 27
  Both | 7 | 12 | 19
  Missing | 36 | 29 | 65
Lumbar radicular pain [Count of Participants; unit: Participants] | 21 | 23 | 44
Previous physiotherapy [Count of Participants; unit: Participants] | 38 | 37 | 75
Previous or scheduled low back surgery [Count of Participants; unit: Participants] | 9 | 6 | 15
Body Mass Index, continuous [Median (Inter-Quartile Range); unit: Kg/m2] | 28.26 [24.05 to 33.34] | 28.30 [23.71 to 31.93] | 28.3 [23.87 to 32.78]
Comorbidities - High Blood Pressure [Count of Participants; unit: Participants] | 23 | 24 | 47
Comorbidities - High Blood Sugar or Diabetes [Count of Participants; unit: Participants] | 8 | 8 | 16
Comorbidities - Cardiac Conditions [Count of Participants; unit: Participants] | 5 | 2 | 7
Comorbidities - Respiratory Conditions [Count of Participants; unit: Participants] | 10 | 10 | 20
Comorbidities - None [Count of Participants; unit: Participants] | 38 | 37 | 75

OUTCOME MEASURES:

1. Primary Outcome: Oswestry Disability Index Score (ODI)
Description: The minimum value of the score is 0% and the maximum is 100%, with lower scores translating into lower disability. In this study, we will be assessing the change between baseline and 8 weeks in Oswestry Disability Index score.
Time Frame: Baseline and 8 weeks after initiation of rehabilitation program
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 70 | 70
units on a scale
  Baseline | 24.84 [19.93 to 28.75] | 25.34 [21.91 to 28.77]
  8-weeks | 17.94 [6.37 to 19.72] | 18.99 [15.20 to 22.78]
  Change baseline-8 weeks | -6.90 [-19.33 to -1.57] | -6.35 [-10.36 to -3.83]
Statistical Analysis 1: Comparison: Digital Rehabilitation vs Conventional Rehabilitation at an Outpatient Clinic; Test type: Equivalence — For a power of 80% and a two-sided 0.05 significance level, we calculated that 102 individuals would be necessary to detect a 10-point difference between the two groups. To guarantee that the study was adequately powered to detect equivalence, a posteriori analysis was conducted using the Two One-Sided Test (TOST) methodology (simulation-based power analysis); p = 0.412, Quantile mixed-effects model — the threshold for statistical significance was set at 0.05; robust method on the medians; Median Difference (Net) = -0.55, 95% CI 2-sided [-2.42 to 5.81]
Statistical Analysis 2: Comparison: Digital Rehabilitation vs Conventional Rehabilitation at an Outpatient Clinic; Test type: Equivalence; p = 0.849, Regression, Logistic — The threshold for statistical analysis was set at 0.05; Odds Ratio (OR) = 0.926, 95% CI 2-sided [0.42 to 2.05]

2. Secondary Outcome: Pain Level
Description: Change in pain level Measured through the following question: "On a scale of 0 to 10, where 0 is no pain and 10 the worst pain imaginable, how would you rate your pain in the last 24 hours?" Minimum and maximum values of the scale are respectively 0 and 10, with lower values representing less pain.
Time Frame: Baseline and 8 weeks after initiation of rehabilitation program
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 70 | 70
units on a scale
  Baseline | 5.40 [4.59 to 6.02] | 5.49 [5.05 to 5.94]
  8-weeks | 3.59 [2.67 to 4.52] | 3.38 [2.71 to 4.05]
  Change baseline-8 weeks | -1.81 [-3.51 to -0.25] | -2.11 [-2.82 to -1.49]
Statistical Analysis 1: Comparison: Digital Rehabilitation vs Conventional Rehabilitation at an Outpatient Clinic; Test type: Equivalence; p = 0.666, Quantile mixed-effects model — The threshold for statistical significance was set at 0.05; robust method on the medians; Median Difference (Net) = 0.30, 95% CI 2-sided [-0.71 to 1.10]

3. Secondary Outcome: Work Productivity and Activity Impairment (WPAI) Overall
Description: Change in WPAI overall scores. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes, with a minimum of 0% and a maximum of 100%.
Time Frame: Baseline and 8 weeks after initiation of rehabilitation program
Population: This analysis includes only participants who completed the WPAI Overall questionnaire. Participants who did not respond to this questionnaire were excluded from the analysis. Consequently, the total number of participants analyzed for this outcome differs from the overall number of participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 45 | 45
units on a scale
  Baseline | 25.61 [13.81 to 30.80] | 23.79 [18.84 to 28.74]
  8-weeks | 16.87 [0.00 to 18.98] | 17.67 [10.29 to 25.05]
  Change baseline-8 weeks | -8.74 [-25.98 to -2.72] | -6.12 [-9.25 to 4.97]
Statistical Analysis 1: Comparison: Digital Rehabilitation vs Conventional Rehabilitation at an Outpatient Clinic; Test type: Equivalence; p = 0.122, Quantile mixed-effects model — The threshold for statistical significance was set at 0.05; Robust test on the medians; Median Difference (Net) = -2.62, 95% CI 2-sided [-14.87 to 4.80]

4. Secondary Outcome: Interest in Undergoing Surgery
Description: Change in surgery intent measured through the following question: "On a scale of 0 to 10, where 0 is not at all and 10 is extremely interested, how interested are you in undergoing back surgery in the next 12 months"? Minimum and maximum values of the scale are respectively 0 and 10, with lower values representing a lower interest.
Time Frame: Baseline and 8 weeks after initiation of rehabilitation program
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 70 | 70
units on a scale
  Baseline | 6.43 [0.00 to 20.68] | 9.76 [4.88 to 14.64]
  8-weeks | 0.06 [0.00 to 1.49] | 0.06 [0.00 to 4.77]
  Change baseline-8 weeks | -6.37 [-25.06 to -2.92] | -9.69 [-13.60 to -4.38]
Statistical Analysis 1: Comparison: Digital Rehabilitation vs Conventional Rehabilitation at an Outpatient Clinic; Test type: Equivalence; p = 0.788, Quantile mixed-effects model — The threshold for statistical significance was set at 0.05; Robust method on the medians; Median Difference (Net) = 3.32, 95% CI 2-sided [-3.11 to 5.90]

5. Secondary Outcome: Medication Consumption
Description: Change in medication consumption, measured through the following questions:
  i. "Are you taking any medication for your low back pain?"; binary score ii. "If yes, are you taking opioids for your low back pain?"; binary score iii. "If yes, on how many days in a week, on average, are you taking medication for your low back pain" minimum 0; max 7 days, with 7 being worse.
Time Frame: Baseline and 8 weeks after initiation of rehabilitation program
Population: This analysis includes only participants who reported medication consumption at baseline. Participants who did not report medication use at baseline were excluded from this analysis. As a result, the total number of participants analyzed for this outcome differs from the overall number of participants enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 34 | 43
Participants | 9 | 7
Statistical Analysis 1: Comparison: Digital Rehabilitation vs Conventional Rehabilitation at an Outpatient Clinic; Test type: Equivalence; p = 0.081, Regression, Logistic — The threshold for statistical significance was set at 0.05; LR to assess the odds between groups for consuming analgesics at 8 weeks using the CG as a reference; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.00 to 1.23]
Statistical Analysis 2: Comparison: Digital Rehabilitation vs Conventional Rehabilitation at an Outpatient Clinic; Test type: Equivalence; p = 0.985, Regression, Logistic — The threshold for statistical significance was set at 0.05; LR to assess the odds between groups for consuming opioids at 8 weeks using the CG as a reference; Odds Ratio (OR) = 0.26, 95% CI 2-sided [0.00 to 1.71]

6. Secondary Outcome: Fear Avoidance Beliefs - Physical Activity (FABQ-PA)
Description: Change in Fear avoidance beliefs-Physical Activity questionnaire - Physical Activity subscale. The questionnaire consists of 4 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 24 and a minimum score of 0. Lower scores mean lower fear avoidance.
Time Frame: Baseline and 8 weeks after initiation of rehabilitation program
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 70 | 70
units on a scale
  Baseline | 14.41 [12.06 to 14.78] | 13.99 [12.50 to 15.48]
  8-weeks | 12.48 [8.41 to 12.71] | 12.48 [10.65 to 14.32]
  Change baseline-8 weeks | -1.92 [-5.48 to 2.48] | -1.50 [-3.28 to 0.03]
Statistical Analysis 1: Comparison: Digital Rehabilitation vs Conventional Rehabilitation at an Outpatient Clinic; Test type: Equivalence; p = 0.871, Quantile mixed-effects model — the threshold for statistical significance was set at 0.05; Robust method on the medians; Median Difference (Net) = -0.42, 95% CI 2-sided [-2.10 to 1.78]

7. Secondary Outcome: Anxiety
Description: Change in the General Anxiety Disorder-7 scale score. Minimum score zero; maximum score 21. Lower scores indicate less severe anxiety.
Time Frame: Baseline and 8 weeks after initiation of rehabilitation program
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 70 | 70
units on a scale
  Baseline | 3.79 [1.32 to 5.88] | 4.22 [2.92 to 5.51]
  8-weeks | 2.51 [0.00 to 2.72] | 2.51 [1.36 to 3.67]
  Change baseline-8 weeks | -1.28 [-4.35 to -0.91] | -1.70 [-2.16 to -0.30]
Statistical Analysis 1: Comparison: Digital Rehabilitation vs Conventional Rehabilitation at an Outpatient Clinic; Test type: Equivalence; p = 0.360, Quantile mixed-effects model — The threshold for statistical significance was set at 0.05; Robust method on the medians; Median Difference (Final Values) = 0.43, 95% CI 2-sided [-0.59 to 1.59]

8. Secondary Outcome: Patient Satisfaction With Intervention
Description: Measured through the following question: "On a scale from 0 to 10, how likely would you recommend this program to a friend or colleague?". Minimum value is zero and maximum is 10. Higher scores translate higher satisfaction.
Time Frame: 8 weeks after initiation of rehabilitation program.
Population: This analysis includes only participants who completed the allocated digital or conventional interventions.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 57 | 45
units on a scale | 8.4 (2.0) | 8.4 (2.6)
Statistical Analysis 1: Comparison: Digital Rehabilitation vs Conventional Rehabilitation at an Outpatient Clinic; Test type: Equivalence; p = 0.837, t-test, 2 sided — The threshold for statistical significance was set at 0.05; Mean Difference (Final Values) = 0.09

9. Secondary Outcome: Physical Activity Levels
Description: Change in the International Physical Activity Questionnaire- Short Form. The scale scores are calculated to provide a qualitative score: low, moderate and high with higher scores translating into higher activity levels.
Time Frame: Baseline and 8 weeks after initiation of rehabilitation program
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 57 | 45
Participants
  Baseline: High | 17 | 14
  Baseline: Moderate | 19 | 16
  Baseline: Low | 21 | 15
  8-weeks: High | 23 | 17
  8-weeks: Moderate | 20 | 15
  8-weeks: Low | 14 | 13
Statistical Analysis 1: Comparison: Digital Rehabilitation vs Conventional Rehabilitation at an Outpatient Clinic; Test type: Equivalence; p = 0.886, Ordinal Regression — The threshold for statistical significance was 0.05; Z-score = -1.28

10. Secondary Outcome: Depression
Description: Change in the Patient Health Questionnaire 9 - 7 scale score. Minimum score zero; maximum score 27. Lower scores indicate less severe depression.
Time Frame: Baseline and 8 weeks after initiation of rehabilitation program
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 70 | 70
units on a scale
  Baseline | 4.09 [0.45 to 4.87] | 4.67 [3.54 to 5.80]
  8-weeks | 3.22 [1.05 to 3.67] | 2.48 [1.44 to 3.52]
  Change baseline-8-weeks | -0.87 [-4.43 to -0.51] | -2.19 [-2.86 to -1.14]
Statistical Analysis 1: Comparison: Digital Rehabilitation vs Conventional Rehabilitation at an Outpatient Clinic; Test type: Equivalence; p = 0.095, Quantile mixed-effects model — The threshold for statistical significance was set at 0.05; Robust method on the medians; Median Difference (Net) = 1.33, 95% CI 2-sided [-2.20 to 2.46]

11. Secondary Outcome: Retention Rate
Description: Number of participants that complete the 8 week program.
Time Frame: Between baseline and 8 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 70 | 70
Participants | 57 | 45

12. Secondary Outcome: Treatment Intensity
Description: Total number of minutes spent doing exercise sessions.
Time Frame: Between baseline and 8 weeks.
Population: This analysis includes only participants who received the allocated intervention. Participants who did not receive the intervention were excluded from this analysis. Therefore, the total number of participants analyzed for this outcome differs from the overall number of participants enrolled in the study.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 63 | 57
minutes | 451.78 (227.36) | 385.98 (145.36)
Statistical Analysis 1: Comparison: Digital Rehabilitation vs Conventional Rehabilitation at an Outpatient Clinic; Test type: Equivalence; p = 0.662, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was set at 0.05; Mean Difference (Final Values) = 65.8

13. Secondary Outcome: Work Productivity and Activity Impairment (WPAI) Work
Description: Change in WPAI work scores. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes, with a minimum of 0% and a maximum of 100%
Time Frame: Baseline and 8 weeks after initiation of rehabilitation program
Population: This analysis includes only participants who completed the WPAI Work questionnaire. Participants who did not respond to this questionnaire were excluded from the analysis. Consequently, the total number of participants analyzed for this outcome differs from the overall number of participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 43 | 44
units on a scale
  Baseline | 23.52 [11.32 to 29.49] | 22.51 [17.62 to 27.40]
  8-weeks | 15.33 [0.00 to 17.62] | 16.29 [8.86 to 23.73]
  Change baseline-8 weeks | -8.19 [-22.87 to 0.03] | -6.22 [-10.14 to 2.68]
Statistical Analysis 1: Comparison: Digital Rehabilitation vs Conventional Rehabilitation at an Outpatient Clinic; Test type: Equivalence; p = 0.246, Quantile mixed-effects model; Robust method on the medians; Median Difference (Net) = -1.97, 95% CI 2-sided [-12.69 to 3.33]

14. Secondary Outcome: Work Productivity and Activity Impairment (WPAI) Time
Description: Change in WPAI time scores. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes, with a minimum of 0% and a maximum of 100%
Time Frame: Baseline and 8 weeks after initiation of rehabilitation program
Population: This analysis includes only participants who completed the WPAI Time questionnaire. Participants who did not respond to this questionnaire were excluded from the analysis. Consequently, the total number of participants analyzed for this outcome differs from the overall number of participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 43 | 44
units on a scale
  Baseline | 3.35 [0.00 to 13.08] | 2.63 [0.29 to 4.96]
  8-weeks | 0.00 [0.00 to 13.08] | 0.00 [0.00 to 2.34]
  Change baseline-8 weeks | -3.36 [-9.01 to -1.51] | -2.63 [-4.38 to -1.99]
Statistical Analysis 1: Comparison: Digital Rehabilitation vs Conventional Rehabilitation at an Outpatient Clinic; Test type: Equivalence; p = 0.408, Quantile mixed-effects model — the threshold for statistical significance was set at 0.05; Robust method on the medians; Median Difference (Net) = -0.73, 95% CI 2-sided [-6.50 to 2.69]

15. Secondary Outcome: Work Productivity and Activity Impairment (WPAI) Activity
Description: Change in WPAI Activity scores. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes, with a minimum of 0% and a maximum of 100%
Time Frame: Baseline and 8 weeks after initiation of rehabilitation program
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 70 | 70
units on a scale
  Baseline | 35.59 [27.39 to 44.10] | 36.73 [29.60 to 43.87]
  8-week | 22.66 [1.11 to 28.34] | 23.45 [17.22 to 29.69]
  Change baseline-8 weeks | -12.93 [-32.09 to -3.11] | -13.28 [-19.27 to -7.38]
Statistical Analysis 1: Comparison: Digital Rehabilitation vs Conventional Rehabilitation at an Outpatient Clinic; Test type: Equivalence; p = 0.650, Quantile mixed-effects model — The threshold for statistical significance was set at 0.05; Robust method on the medians; Median Difference (Net) = 0.35, 95% CI 2-sided [-6.22 to 9.87]

16. Secondary Outcome: Dropout Rate
Description: Rate of patients who dropout from the program
Time Frame: Program-end
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 70 | 70
Participants | 11 | 24
Statistical Analysis 1: Comparison: Digital Rehabilitation vs Conventional Rehabilitation at an Outpatient Clinic; Test type: Equivalence; p = 0.019, Chi-squared; Difference in proportions = 18.6

17. Secondary Outcome: Total Sessions
Description: Number of sessions performed at program-end
Time Frame: 8 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 63 | 57
sessions | 22.32 (9.46) | 12.42 (4.95)

18. Secondary Outcome: Frequency of Sessions Per Week
Description: Number of sessions performed per week in the 8-week rehabilitation program
Time Frame: 8-weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: sessions per week
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
Number analyzed (Participants) | 63 | 57
sessions per week | 2.79 (1.18) | 1.55 (0.62)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: The total number of participants at risk for adverse events differs from the overall number of participants enrolled in the study, as only participants who received the allocated interventions were considered.
  Both participants and physical therapists were instructed to contact the study investigators when adverse events occurred (registered on Castor Electronic Data Capture).
Arm/Group | Digital Rehabilitation | Conventional Rehabilitation at an Outpatient Clinic
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/57
Other Adverse Events (participants affected / at risk) | 11/63 | 6/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digital Rehabilitation (N=63) | Conventional Rehabilitation at an Outpatient Clinic (N=57)
Brain Bleeding (Vascular disorders) | 1 (1) | 0 (0) — Not related to Study Intervention. Severity: Severe. Action taken with study treatment: None.
Spine Procedure (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Lumbar medial branch block. Unlikely related to Study Intervention. Severity: Moderate. Action taken with study treatment: Other.
Chest Pain (General disorders) | 1 (1) | 0 (0) — Development of Chest Pain with visit to emergency room. Not related to Study Intervention. Severity: Moderate. Action taken with study treatment: None.
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) — Not related or unlikely related to Study Intervention. Severity: Mild. Action taken with study treatment: None, Intervention discontinued, or Change of treatment program.
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unlikely related to Study Intervention. Severity: Moderate. Action taken with study treatment: None.
Covid-19 infection (Infections and infestations) | 1 (1) | 0 (0) — Not related to Study Intervention. Severity: Mild. Action taken with study treatment: Change of treatment program.
Low Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) — Worsening pain or injury after moving. Not related or unlikely related to Study Intervention. Severity: Mild or Moderate. Action taken with study treatment: None, Change of treatment program, or Other.
Arm Cyst (Infections and infestations) | 1 (1) | 0 (0) — Urgent care needed. Not related to Study Intervention. Severity: Mild. Action taken with study treatment: Other.
Foot Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Not related to Study Intervention. Severity: Mild. Action taken with study treatment: Other.
Lumbar Spinal Injection Reaction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Not related to Study Intervention. Severity: Moderate. Action taken with study treatment: Change of treatment program.
Ankle Sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Not related to Study Intervention. Severity: Mild. Action taken with study treatment: None.
Struck by Car (Social circumstances) | 0 (0) | 1 (1) — Not related to Study Intervention. Severity: Moderate. Action taken with study treatment: Change of treatment program.
Cold sickness (Infections and infestations) | 0 (0) | 1 (1) — Not related to Study Intervention. Severity: Mild. Action taken with study treatment: None.

LIMITATIONS AND CAVEATS:
Lack of (i) blinding of patients, physical therapists, and investigators due to the intervention's nature; (ii) objective outcome measures (eg, muscle strength, range of motion); (iii) an externally blinded outcome adjudicator. The COVID-19 pandemic may have positively influenced compliance. Higher dropout in the conventional group highlights the need for strategies like additional contacts. Greater granularity in pharmacological data (type, dosage, frequency) is necessary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT04808141/Prot_SAP_ICF_000.pdf